CLINICAL TRIAL: NCT06161870
Title: Clinical Study of Individualized Vancomycin Dosing Based on Population Pharmacokinetic Model for Severe Infections
Brief Title: Clinical Study of Individualized Vancomycin Dosing Based on Population PK Model
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Hainan Zhang, Director of the neurology department, Central South University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021SK53501
Record Dates: First submitted 2023-10-24; First posted 2023-12-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-11

CONDITIONS: Severe Infection
Keywords: vancomycin; population pharmacokinetic model; severe infection
MeSH Terms: conditions — Infections | interventions — Models, Biological

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- experimental group (Experimental): The experimental group will be guided by the population pharmacokinetics (PK) model for individual dosing of vancomycin.
  Interventions: Drug: individualized vancomycin dosing based on the population pharmacokinetics (PK) model
- control group (Other): The control group will be administered empirically (15-20 mg/kg vancomycin infused intermittently every 8-12 hours depending on the actual body weight of participants).
  Interventions: Drug: empirical vancomycin dosing

INTERVENTIONS:
Drug: individualized vancomycin dosing based on the population pharmacokinetics (PK) model — The experimental group will be guided at the bedside with individualized vancomycin dosing by a drug dosimetry software tool that incorporates a PK model developed by Roberts JA et al. for data from sepsis patients. The model developed by Roberts JA et al. has been validated in multiple centers to have a good ability to predict the concentration-time data of patients. Once the basic information of participants such as gender, age, body weight, and creatinine clearance rate (CCR) is entered, the software tool can calculate the dosing regimen that is estimated to achieve the pharmacodynamic (PD) target. The area under the curve (AUC24) of 400-600mg·h/L is identified as the PD target of vancomycin.
  Arms: experimental group
Drug: empirical vancomycin dosing — The control group will be administered empirically (15-20 mg/kg vancomycin infused intermittently every 8-12 hours depending on the actual body weight of participants).
  Arms: control group

SUMMARY:
The goal of this clinical trial is to compare the clinical efficacy of individualized dosing based on the population pharmacokinetics (PK) model and empirical dosing of vancomycin in participants with severe infections.

It aims to answer whether individual vancomycin dosing based on population PK model is superior to empirical dosing in terms of clinical efficacy and safety.

Participants will be randomly divided into experimental group and control group. The experimental group will be guided by the population PK model for individual dosing, and the control group will be given empirical dosing. Demographic data, clinical characteristics of participants, and their trough concentrations (Cmin) and peak concentrations (Cmax) of vancomycin will be collected. Area under the concentration curve (AUC24) of participants will be calculated using the first-order PK equation.

Researchers will compare experimental group and control group to see if individual vancomycin dosing based on population PK model is superior to empirical dosing in terms of clinical efficacy and safety.

DETAILED DESCRIPTION:
1. Research purpose The goal of this clinical trial is to compare the clinical efficacy of individualized dosing based on the population pharmacokinetics (PK) model and empirical dosing of vancomycin in participants with severe infections.

   It aims to answer whether individual vancomycin dosing based on population PK model is superior to empirical dosing in terms of clinical efficacy and safety.
2. Research methods 112 subjects who are treated with vancomycin for severe infections caused by suspected or confirmed gram-positive cocci during hospitalization in the Second Xiangya Hospital of Central South University will be prospectively collected (sample size is calculated according to the sample size calculation formula for clinical trials of merits and demerits). Severe gram-positive infection is defined in this study as bacteremia, sepsis, infective endocarditis, pneumonia, and encephalitis/meningitis caused by gram-positive infection with clinical suspicion or evidence of microbiological culture. Eligible participants will be screened according to the inclusion and exclusion criteria established in this study. All excluded cases should be recorded for future reference. At the end of the test, the shedding rate will be calculated and the safety analysis will be carried out.

   Before the implementation of the study, the research designer will use computer programmed data processing to generate a random sequence, and the group of participants will be determined according to random numbers. Participants will be randomly assigned to the experimental group and the control group. A single-blind method will be used. Study designers, clinicians, and statistical analysts will be aware of groups of participants, but they do not disclose this information to participants or their authorized representatives.

   The experimental group will be guided at the bedside with individualized vancomycin dosing by a drug dosimetry software tool that incorporates a PK model developed by Roberts JA et al. for data from sepsis patients. The model developed by Roberts JA et al. has been validated in multiple centers to have a good ability to predict the concentration-time data of patients. Once the basic information of participants such as gender, age, body weight, and creatinine clearance rate (CCR) is entered, the software tool can calculate the dosing regimen that is estimated to achieve the pharmacodynamic (PD) target. The area under the curve (AUC24) of 400-600mg·h/L is identified as the PD target of vancomycin. The control group will be administered empirically (15-20 mg/kg vancomycin infused intermittently every 8-12 hours depending on the actual body weight of participants).

   The trough concentration (Cmin) and peak concentration (Cmax) of vancomycin in the two groups will be measured after the dosing of vancomycin achieve steady state, and the CCR, volume of distribution (Vd) and AUC24 of vancomycin will be calculated based on the first-order PK equation. In addition, demographic data and clinical data of both groups of participants will be collected. Demographic data included sex, age, height, body weight, and body mass index（BMI）. Clinical data included serum creatinine（SCR）, CCR, serum albumin level, vancomycin dosage regimen, body temperature, white blood cell count (WBC), percentage of neutrophils (NEUT%), serum procalcitonin (PCT), serum C-reactive protein (CRP), Acute physiology and Chronic Health Evaluation (APACHE) Ⅱ, Sequential Organ Failure Assessment (SOFA), length of neurological intensive care unit (NICU) stay, 30-day outcomes, and 90-day outcomes. In addition, vancomycin-related adverse reactions and the use of concomitant nephrotoxic drugs will also be collected.

   The vancomycin concentrations, demographic data, and clinical data of the two groups of participants will be recorded in the case report forms.

   Vancomycin concentrations and clinical data collected after the end of vancomycin treatment will be compared between the two groups to answer whether individualized vancomycin dosing based on population PK model is superior to empirical treatment in terms of clinical efficacy and safety.
3. Statistics analysis method SPSS 26.0 software will be used for statistical analysis. Independent sample t test or Mann-Whitney U test in non-parametric test will be used for comparison of continuous data between groups. Chi-square test is used for comparison of nominal data between groups. All tests are two-tailed, and p < 0.05 is considered statistically significant.
4. Data processing and Record preservation 4.1 Preservation of case report forms Based on the original data of the participants, the investigator will record the data in the case report form in a timely, complete, correct and true manner. The investigator will confirm that all case report forms are correctly completed and consistent with the original data. The case report form should be signed by the operator and the reviewer. Any errors and omissions should be corrected in a timely manner. The original records should be kept clear and visible during the modification, and the modification should be signed and dated by the researcher.

4.2 Data collection, entry and management All original records should be filled in carefully according to the protocol, and any corrections should be underlined. Marginalization of corrected data should be signed and dated by the investigator and should not erase or overwrite the original records. Before data entry, understand the content of each item recorded. Database naming should be standardized, legible, and easy to find. The investigator should ensure its accuracy, safety and confidentiality. After the data entry, the data in some records should be checked to understand the quality of the input, and the existing problems should be analyzed and solved. After the completion of the study, the statisticians should further confirm that the selected samples fully meet the requirements of the inclusion criteria according to the inclusion criteria specified in the protocol, and carefully verify whether there are samples that meet the exclusion criteria. If there are, they should be removed during the statistics, and the reasons for exclusion should be described in the report. All samples that meet the requirements of the study will be statistically analyzed according to the statistical methods specified in the protocol. The statistical data and results will be faithfully recorded and provided to the report writer for report preparation.

ELIGIBILITY:
Inclusion Criteria:

1. Admission to neurological intensive care unit (NICU).
2. Age ≥18 years old. Participants will be eligible if they meet both of these criteria.

Exclusion Criteria:

1. Evidence of absolute renal impairment, which included Serum creatinine (SCR) ≥133 μmol/L at admission, development of acute kidney injury (AKI) after admission, need for renal replacement therapy during hospitalization, renal related tests suggestive of renal disease, and previous history of renal replacement therapy or chronic kidney disease.
2. Pregnant participants.
3. Primary diagnosis is non-neurological disease.
4. The height or weight of participants is not recorded in the medical record system.
5. The frequency of SCR monitoring was less than 3 times. Participants who meet any of these criteria will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Area under the Plasma Concentration versus Time Curve within 24 hours (AUC24) of vancomycin | Half an hour before the fourth dose, and 1 hour after the end of the fourth dose
  After three consecutive doses of vancomycin, trough concentration (Cmin) will be measured by blood sampling half an hour before the fourth dose, and peak concentration (Cmax) will be measured by blood sampling 1 hour after the end of the fourth dose to calculate AUC24.

SECONDARY OUTCOMES:
Mean scores of Acute Physiology and Chronic Health Evaluation (APACHE)Ⅱ after 2 weeks of vancomycin treatment | After 2 weeks of vancomycin treatment
  After 2 weeks of vancomycin treatment, APACHEⅡ of each participant will be collected to calculate mean scores.
Mean scores of Sequential Organ Failure Assessment (SOFA) after 2 weeks of vancomycin treatment | After 2 weeks of vancomycin treatment
  After 2 weeks of vancomycin treatment, SOFA of each participant will be collected to calculate mean scores.
Survival status (alive or dead) of participants at day 30 of hospitalization | Day 30 of hospitalization
  The survival status (alive or dead) of each participant will be recorded at day 30 of hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Hainan Zhang, Doctor, Principal Investigator — Central South University
Locations (1):
- Central South University, Changsha, Hunan, China